CLINICAL TRIAL: NCT03609138
Title: The O-arm Assessment of Vertebral Movement Pre and Post Correction Using ST2R Technique
Brief Title: O-arm Assessment of Vertebral Movement Using ST2R Technique
Status: Withdrawn | Type: Observational
Why Stopped: Study aborted
Sponsor: Medicrea, USA Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: #0312
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Study Cohort
  Interventions: Device: Spinal Hardware

INTERVENTIONS:
Device: Spinal Hardware — Pedicle screws and patient specific rods

SUMMARY:
The study is quantifying how the patients' back has been corrected using Medicrea's hardware through imaging taken before,during and after the surgery.

DETAILED DESCRIPTION:
Visits include the pre-operative visit, 1 and 2 year follow-up visits. Participation includes answering questions and filling out questionnaires. There are no immediate benefits by joining this study, but could potentially help define better techniques for the future spine surgeries. The risks involved in this study are minimal and there are no alternatives to this study.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent idiopathic scoliosis requiring selective thoracic posterior spinal instrumentation and fusion with the PASS LP system (screws, rods, hooks) and UNiD rod technology
* Age between 10 and 21
* Lenke Type 1 curve
* Consent and Assent to participate in the study

Exclusion Criteria:

* Age superior to 21 years
* Spinal deformities other than Lenke 1 type
* Use of implant other than those from the PASS LP system or sublaminar bands
* Neuromuscular or degenerative scoliosis
* Spinal cord abnormalities with any neurologic symptoms or signs
* Spinal cord lesions requiring neurosurgical interventions, such as hydromyelia requiring Arnold Chiari decompression
* Primary muscle diseases (e.g. Charcot-Marie Tooth, Guillain-Barre syndrome, Cerebral palsy, or Spina bidifa, Neurofibroma)
* Primary abnormalities of bones (e.g. osteogenesis imperfect)
* Congenital Scoliosis
* Scoliosis requiring anterior release
* Previous spinal surgery
* Absence of required preoperative data (diagnosis, consent…)

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients diagnosed with adolescent idiopathic scoliosis undergoing fusion surgery
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Quantify vertebral derotation with ST2R technique in AIS for Lenke Type 1 patients | 4 years

SECONDARY OUTCOMES:
Assess 3 dimensional correction pre- and post- correction using x-rays and O-arm data | 4 years

IPD SHARING:
Plan to Share IPD: Undecided